CLINICAL TRIAL: NCT05587647
Title: The Effect of Transition to Adulthood Education Program Given to Mothers of Children With Intellectual Disability on Family Quality of Life and Perceived Stress Level
Brief Title: The Effect of Transition to Adulthood Education Program on Family Quality of Life and Perceived Stress Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Eysan Hanzade Umac, Teaching and Research Assistant, Koç University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Eyşan Umac
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Intellectual Disability
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: YEGEP group/Intervention (Experimental): Mothers will be informed about the program and invited to work. In the phone call, information will be given about the purpose, duration, requirements and volunteering of the study. The planned training schedule will be applied to these mothers.
  Interventions: Other: Transition to Adulthood Education Program
- Control group (No Intervention): Annual care trainings are given to parents at the disabled center where the study will be conducted. There is no similar practice to these mothers on the same dates. place in the control group

INTERVENTIONS:
Other: Transition to Adulthood Education Program — YEGEP was developed by the authors based on the information in the literature, based on the needs of mothers of children who have reached adulthood or are going through. Three training modules are planned in line with current requirements. Education will also be supported by audio-visual and written materials. It is planned that the trainings, which will last for 3 weeks in total, for 1 hour a week for each group, in the form of 3 sessions of 1 hour with these contents, will be held at a disabled center. Titles of training modules:
  1. Developmental Period Characteristics of Young Adults with Intellectual Disabilities (Transition to Adulthood, Future Planning / Social Life (employment, peers, etc.)
  2. Protecting and Sustaining the Health of Young Adult with Intellectual Disabilities
  3. Coping with Stress
  Other Names: There is no other intervention
  Arms: Experimental: YEGEP group/Intervention

SUMMARY:
Negative emotions experienced during life processes and the burden of caregiving affect the quality of life of parents. It has been found that parents who care for their children with intellectual disability (ID) for a long time have difficulties in coping with stress and their quality of life is adversely affected. However, families play a key role in maintaining the care of their children with ID, so it is very important that parents are supported in the matters they need.

DETAILED DESCRIPTION:
Mothers are generally the people who take on a large part of the burden of care for their children with intellectual disability (ID) in the family and are most affected by the negativities brought by the conditions. Providing support to mothers for the care and future planning of their children who have just passed into adult life and for their future planning is important both in terms of maintaining family well-being and creating positive effects in the lives of individuals with mental disabilities.

With this study, it is aimed to increase the quality of life of mothers and to reduce perceived stress levels with the training (YEGEP) modules to be given for the changing care needs of individuals with ID who have reached adulthood or are in transition. In addition, it is expected that the health risks of young adults with ID will be determined at an early stage, and their health will be improved and protected.

ELIGIBILITY:
Inclusion Criteria:

* Whose child is registered with the disability center,
* Have a young adult child between the ages of 20 and 35 with moderate and severe mental disabilities,
* Speaking Turkish and literate Turkish,
* Not visually and speech impaired,
* Mothers who volunteered to participate in the study will be included.

Exclusion Criteria:

• Mothers who did not volunteer to participate in the study and were illiterate in Turkish were not included in the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | All mothers will be asked to fill in 1 hour before the training.
  The personal information form consists of various socio-demographic questions about the participant and the mentally handicapped child, such as gender, age and educational status.
Beach Center Family Quality of Life (BCFQOL) Scale | Immediately after the training is completed (average of 5 minutes), mothers will be asked to complete this scale.
  The scale, developed by University of Kansas Beach Center on Family and Disability (2006) (Beach Center on Disability at the University of Kansas in partnership with families, 2006) and adapted into Turkish by Meral et al. (2012), consists of 25 questions, five sub-dimensions and 5 It is a data collection tool consisting of likert-type responses. The scale aims to determine the quality of life of families with children with special needs.
Beach Center Family Quality of Life (BCFQOL) Scale | One month after the training is completed, mothers will be asked to complete this scale to evaluate the effectiveness of the training.
  The scale, developed by University of Kansas Beach Center on Family and Disability (2006) (Beach Center on Disability at the University of Kansas in partnership with families, 2006) and adapted into Turkish by Meral et al. (2012), consists of 25 questions, five sub-dimensions and 5 It is a data collection tool consisting of likert-type responses. The scale aims to determine the quality of life of families with children with special needs.
Perceived Stress Scale | Immediately after the training is completed (average of 5 minutes), mothers will be asked to complete this scale.
  The scale developed by Cohen, Kamarck, and Mermelstein (1983) to measure how individuals evaluate stressful life events as unpredictable, uncontrollable and difficult to cope with in the last month consists of 10 items.
Perceived Stress Scale | Immediately afteImmediately after the training is completed (average of 5 minutes), mothers will be asked to complete this scale.r the training is completed (average of 5 minutes), mothers will be asked to complete this scale.
  The scale developed by Cohen, Kamarck, and Mermelstein (1983) to measure how individuals evaluate stressful life events as unpredictable, uncontrollable and difficult to cope with in the last month consists of 10 items.

CONTACTS AND LOCATIONS:
Locations (1):
- Koc University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No